CLINICAL TRIAL: NCT02284256
Title: A Phase 3b, Randomized, Single-Blind, Controlled, Comparative Efficacy and Safety Study of Topical FibrocapsTM (RaplixaTM) and Tachosil® in Surgical Hemostasis During Hepatic Resection
Brief Title: A Safety and Efficacy Study Comparing Fibrocaps and Tachosil in Hepatic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FC-005; 2014-000816-32 (EudraCT Number)
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Surgical Bleeding
MeSH Terms: interventions — Fibrin Tissue Adhesive; TachoSil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fibrocaps (Experimental): Human fibrinogen and thrombin powder. Single application during surgery
  Other Names:
  * Raplixa
  * PRO-0601
  * Fibrin sealant
  Device: Gelatin sponge. Single application during surgery
  Other Name: Spongostan
  Interventions: Drug: Fibrocaps
- TachoSil (Active Comparator): Human fibrinogen and thrombin powder. Single application during surgery
  Interventions: Drug: TachoSil

INTERVENTIONS:
Drug: Fibrocaps
  Other Names: Raplixa
  Arms: Fibrocaps
Drug: TachoSil
  Arms: TachoSil

SUMMARY:
The primary objective of the study is to demonstrate the non-inferiority or superiority of Fibrocaps plus gelatin sponge compared to Tachosil when control of mild to moderate bleeding with conventional surgical techniques is ineffective or impractical.

ELIGIBILITY:
Inclusion Criteria (pre-surgery):

1. Subject has signed an independent ethics committee (IEC)-approved informed consent document
2. Subject is undergoing hepatic wedge resection or anatomic resection of 1 to 5 contiguous hepatic segments, and/or other hepatic surgery, any of which may be combined with other surgical procedures involving the gall bladder or intestines
3. Subject age is >18 years at time of consent
4. If female and of child-bearing potential, subject has negative pregnancy test during screening and is not breast-feeding
5. If subject is a sexually active male or a sexually active female of child-bearing potential, subject agrees to use a medically accepted form of contraception from the time of consent to completion of all follow-up study visits

   Inclusion Criteria (during surgery):
6. Presence of mild to moderate bleeding/oozing when control by conventional surgical techniques, including but not limited to suture, ligature and cautery is ineffective or impractical
7. Absence of intra-operative complications other than bleeding which, in the opinion of the investigator, may interfere with the assessment of efficacy or safety
8. Approximate TBS surface area of ≤ 100 cm^2

Exclusion Criteria:

1. Subject has known hypersensitivity to Fibrocaps or any of its components
2. Subject has known allergy to porcine gelatin
3. Subject has known hypersensitivity to Tachosil or any of the excipients included in Tachosil
4. Subject is unwilling to receive blood products
5. Subject is having hepatic surgery due to emergency-traumatic event
6. Subject requires extrahepatic bile duct resection (common bile duct resection or resection of the bile duct which leads to performing an anastomoses between the bile duct and small bowel) and biliary anastomosis, and/or pancreatic resections
7. Subject has any clinically-significant coagulation disorder that may interfere with the assessment of efficacy or pose a safety risk to the subject according to the investigator, or baseline abnormalities of international normalized ratio (INR) > 2.5 or activated partial thromboplastin time (aPTT) > 100 seconds during screening that are not explained by current drug treatment (e.g., warfarin, heparin)
8. Subject has a platelet count < 100 x10^9 PLT/L during screening
9. Subject has medical, social or psychosocial factors that, in the opinion of the investigator, could impact safety or compliance with study procedures
10. Subject is currently participating or has participated in another clinical study involving another investigational agent within 4 weeks of the planned date of surgery or is planning participation in another clinical trial within 6 weeks after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Time to Hemostasis (TTH) | Within 5 minutes of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wolf Bechstein, MD, Principal Investigator — J.W.Goethe-Universität; Martin Bodingbauer, MD, Principal Investigator — Medical University of Vienna
Locations (15):
- Austria (3):
  - Universitaetsklinik Innsbruck, Innsbruck
  - Krankenhaus der Barmherzigen Schwestern Linz Betriebsgesellschaft m.b.H., Linz
  - Medizinische Universitaet Wien AKH, Vienna
- Germany (12):
  - Universitaetsklinikum Aachen, RWTH, Aachen
  - Charite Campus Virchow-Klinikum, Berlin
  - Krankenhaus Nordwest GmbH, Frankfurt am Main
  - J. W. Goethe Universitaetsklinik Frankfurt, Frankfurt am Main
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Leipzig AoeR, Leipzig
  - Klinikum Rechts der Isar Munich, Munich
  - Klinikum der LMU Muenchen - Campus Grosshadern, München
  - Klinikum Stuttgart - Katharinenhospital (KH), Stuttgart
  - Universitaetsklinikum Tuebingen, Tübingen